CLINICAL TRIAL: NCT02454179
Title: A Phase 2 Proof-of-Concept Study of the Combination of ACP-196 and Pembrolizumab in Subjects With Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Study of the Combination of Acalabrutinib (ACP-196) and Pembrolizumab in Advanced Head and Neck Squamous Cell Carcinoma
Acronym: KEYNOTE147
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-006
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): pembrolizumab
  Interventions: Drug: pembrolizumab
- Arm 2 (Experimental): acalabrutinib in combination with pembrolizumab
  Interventions: Drug: pembrolizumab; Drug: Acalabrutinib

INTERVENTIONS:
Drug: pembrolizumab
  Other Names: Keytruda
Drug: Acalabrutinib
  Other Names: ACP-196
  Arms: Arm 2

SUMMARY:
Study of the combination of acalabrutinib (ACP-196) and pembrolizumab in subjects with advanced head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Histologically or cytologically confirmed recurrent, metastatic or unresectable HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx that that has either progressed during or after platinum-based chemotherapy administered for metastatic disease or has recurred during or within 6 months after the completion of platinum-based neoadjuvant or adjuvant therapy
* Presence of radiographically measurable disease as defined by RECIST 1.1
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Prior malignancy (other than HNSCC), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years
* Known central nervous system metastases and/or carcinomatous meningitis
* A life-threatening illness, medical condition (including psychiatric conditions) or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of starting study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mono Therapy of Pembrolizumab Arm 1: Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
- Combo Therapy Acalabrutinib + Pembrolizumab Arm 2: Acalabrutinib 100mg PO BID plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Mono Therapy of Pembrolizumab Arm 1 | Combo Therapy Acalabrutinib + Pembrolizumab Arm 2
Started | 39 | 39
Enrolled | 39 | 39
Received Study Medication | 39 | 37
Discontinue Study | 39 | 39
Completed | 0 | 0
Not Completed | 39 | 39

BASELINE CHARACTERISTICS:
Groups:
- Mono Therapy Arm - Pembrolizumab: Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
- Combo Therapy Arm - Acalabrutinib + Pembrolizumab: Acalabrutinib 100mg PO BID plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
- Total: Total of all reporting groups
Arm/Group | Mono Therapy Arm - Pembrolizumab | Combo Therapy Arm - Acalabrutinib + Pembrolizumab | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (10.45) | 61.4 (11.12) | 61.8 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 34 | 35 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 6 | 6
  White | 37 | 29 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 52 weeks
Population: The study participants had to have a minimum of one scan (for tumor assessment) after randomization/treatment in order to be considered analyzed.
  And some of the participants didn't make it to Wk 7 of treatment, hence reduction in the number of subjects analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Combo Therapy Arm - Acalabrutinib and Pembrolizumab: Acalabrutinib 100mg PO BID plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W).
Arm/Group | Mono Therapy Arm - Pembrolizumab | Combo Therapy Arm - Acalabrutinib and Pembrolizumab
Number analyzed (Participants) | 37 | 30
Participants | 7 | 5

ADVERSE EVENTS:
Time Frame: Safety Analysis tracked from 0 day to 2 years.
Groups:
- Arm 1 - Pembrolizumab: Pembrolizumab Monotherapy
- Arm 2 - Acalabrutinib + Pembrolizumab: Acalabrutinib in combination with Pembrolizumab
Arm/Group | Arm 1 - Pembrolizumab | Arm 2 - Acalabrutinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 26/39 | 23/37
Serious Adverse Events (participants affected / at risk) | 12/39 | 25/37
Other Adverse Events (participants affected / at risk) | 39/39 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Pembrolizumab (N=39) | Arm 2 - Acalabrutinib + Pembrolizumab (N=37)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Pulseless Electrical Activity (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Mouth Heamorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2 — General disorders and administration site conditions.
Chest Pain (General disorders) | 1 | 0 — General disorders and administration site conditions.
Urosepsis (Infections and infestations) | 0 | 2
Clostridia Sepsis (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Epiglottistis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour Heaorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypnoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Aneurysm (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthrostatic Hypotension (Vascular disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions
Oedema (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions
Oedema Peripheral (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Sepsis (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Pembrolizumab (N=39) | Arm 2 - Acalabrutinib + Pembrolizumab (N=37)
Mucosal Inflammation (General disorders) | 0 | 2 — General Disorders and administration site conditions.
Oedema (General disorders) | 0 | 2 — General Disorders and administration site conditions.
Seasonal Allergy (Immune system disorders) | 2 | 0
Pneumonia (Infections and infestations) | 4 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 6
Candida Infection (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 1 | 4
Urinary Tract Infection (Infections and infestations) | 3 | 0
Aptyalism (Gastrointestinal disorders) | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 20 | 14 — General Disorders and administration site conditions.
Oedema Peripheral (General disorders) | 4 | 9 — General Disorders and administration site conditions.
Pyrexia (General disorders) | 5 | 8 — General Disorders and administration site conditions.
Asthenia (General disorders) | 2 | 7 — General Disorders and administration site conditions.
Non-Cardiac Chest Pain (General disorders) | 2 | 1 — General Disorders and administration site conditions.
Chills (General disorders) | 2 | 1 — General Disorders and administration site conditions.
Vomiting (Gastrointestinal disorders) | 5 | 7
Dysphagia (Gastrointestinal disorders) | 3 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 3
Oral Pain (Gastrointestinal disorders) | 3 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 12
Tachycardia (Cardiac disorders) | 2 | 2
Sinus Tachycardia (Cardiac disorders) | 0 | 3
Hypothyroidism (Endocrine disorders) | 4 | 2
Vision Blurred (Eye disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 9
Diarrhea (Gastrointestinal disorders) | 6 | 11
Constipation (Gastrointestinal disorders) | 5 | 8
White Blood Cell Count Decreased (Investigations) | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 11
Dehydration (Metabolism and nutrition disorders) | 2 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1
Oral Candidiasis (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Weight Decreased (Investigations) | 5 | 9
Blood Creatinine Increased (Investigations) | 2 | 6
Alanine Aminotransferase Increased (Investigations) | 0 | 4
Aspartate Aminotransferase Increased (Investigations) | 0 | 4
Platelet Count Decreased (Investigations) | 1 | 2
Musculoskeletel Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Headache (Nervous system disorders) | 8 | 7
Dizziness (Nervous system disorders) | 2 | 6
Speech Disorder (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 8
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 2
Eating Disorder (Psychiatric disorders) | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 3
Nocturia (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 7 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 4
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 3
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 5 | 6
Hypertension (Vascular disorders) | 3 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT02454179/SAP_000.pdf
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT02454179/Prot_001.pdf